CLINICAL TRIAL: NCT06998329
Title: PANDORA: PulmonAry hyperteNsion DiagnOsis: a National cohoRt reseArch
Brief Title: PulmonAry hyperteNsion DiagnOsis: a National cohoRt reseArch
Acronym: PANDORA
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Caio Júlio César dos Santos Fernandes, Principal Investigator, University of Sao Paulo General Hospital
Other Study IDs: SGP26817
Record Dates: First submitted 2025-05-13; First posted 2025-05-31 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension (PAH); Pulmonary Arterial Hypertension (PAH) (WHO Group 1 PH); Pulmonary Arterial Hypertension
Keywords: Pulmonary Hypertension; Diagnostic Delay; Right Heart Catheterization; Early Diagnosis; Diagnostic Journey; Risk Stratification; Differential Diagnoses
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Pulmonary Arterial Hypertension: This group includes adult patients diagnosed with Group 1 pulmonary arterial hypertension (PAH), according to international hemodynamic criteria confirmed by right heart catheterization. All patients were diagnosed within the past five years and are followed at participating reference centers in Brazil. This is a non-interventional, observational study based on retrospective and/or prospective data from medical records. No treatment or diagnostic procedure will be administered as part of the study.
  Interventions: Other: There will be no intervention

INTERVENTIONS:
Other: There will be no intervention — There will be no intervention

SUMMARY:
Understanding Delays in the Diagnosis of Pulmonary Arterial Hypertension and Rare Diseases in Brazil: A Multicenter Observational Study

--- Pulmonary arterial hypertension (PAH) is a rare, progressive, and life-threatening disease that affects the arteries of the lungs and the right side of the heart. Early diagnosis is essential to initiate appropriate treatment and improve patient outcomes. However, worldwide studies show that there is often a significant delay between the onset of symptoms and the final diagnosis. This delay may lead to disease progression and worse survival.

This multicenter observational study aims to understand the time from the first symptoms to the diagnosis of PAH and other rare diseases across several Brazilian reference centers. By analyzing medical records and patient journeys, the investigators intends to identify factors contributing to delayed diagnosis and potential opportunities for earlier detection.

The study includes adult patients diagnosed with PAH or other selected rare diseases within the last five years. The investigators will analyze time to diagnosis, number and type of physicians consulted, tests performed, and possible misdiagnoses. Our goal is to support the development of strategies that reduce diagnostic delay and improve access to specialized care for people living with rare diseases.

This study does not involve any intervention and poses no additional risk to participants, as it is based solely on retrospective data from medical records.

DETAILED DESCRIPTION:
Background and Rationale:

Pulmonary arterial hypertension (PAH) is a rare condition characterized by progressive elevation of pulmonary artery pressure, leading to right ventricular dysfunction and death if untreated. Despite advances in therapy and increasing awareness, several studies have consistently shown substantial diagnostic delays. For example, in the Australian DELAY study, the mean time from symptom onset to diagnosis of idiopathic PAH was nearly 4 years (47 ± 34 months), and patients typically visited multiple general practitioners and specialists before referral to a PAH center. In Latin America, similar findings were reported, with patients waiting an average of 1.6 years from first symptoms to diagnosis and over 50% receiving a misdiagnosis, such as asthma or heart failure, prior to PAH confirmation .

Delays are not limited to PAH. For many rare diseases, such as primary immunodeficiencies, sarcoidosis, and myositis, patients often experience a prolonged and complex journey to diagnosis. A recent qualitative study in Australia highlighted delays ranging from months to decades, with barriers including misattribution of symptoms, clinician bias, and fragmentation of care.

In Brazil, data on time to diagnosis for PAH and other rare diseases are limited. Understanding the diagnostic trajectory in the local context is critical to guide health policies and professional education.

Objectives:

The primary objective of this study is to characterize the time from symptom onset to confirmed diagnosis in patients with PAH and other selected rare diseases, and to identify common barriers and facilitators to diagnosis.

Specific Aims:

* Estimate the average and median time from first symptom to diagnosis.
* Quantify the number and types of healthcare professionals consulted before diagnosis.
* Identify common misdiagnoses prior to the final diagnosis.
* Evaluate use and timing of diagnostic tools (e.g., echocardiogram, right heart catheterization, imaging).
* Compare diagnostic delays across regions and reference centers.
* Identify associations between patient characteristics (age, sex, location) and time to diagnosis.

Study Design:

This is a retrospective, multicenter, observational study involving data collection from medical records of patients diagnosed with PAH or other rare diseases in participating reference centers across Brazil. The study will include patients diagnosed in the last five years and will not involve any direct patient contact or intervention.

Participating Centers:

Tertiary hospitals with dedicated outpatient clinics for pulmonary hypertension and rare diseases in major Brazilian cities, including São Paulo, Rio de Janeiro, Recife, Fortaleza, Belém, Vitória, and Curitiba.

Eligibility Criteria:

- Adult patients (≥18 years) diagnosed with PAH (Group 1 PH) or other selected rare diseases.

Confirmed diagnosis based on international or national diagnostic criteria.

- Sufficient medical record data available to estimate time from first symptom to diagnosis.

Data Collection and Analysis:

Data will be extracted from patient records using a standardized case report form. Key variables include:

* Date of symptom onset (as described by patient or noted in clinical notes)
* Date of first medical consultation
* Number of general practitioner and specialist visits before diagnosis
* Diagnostic tests performed and their dates
* Initial diagnoses prior to final diagnosis
* Date of confirmed diagnosis (e.g., date of right heart catheterization in PAH)
* Demographic information (age, sex, region, referral source)

Quantitative analyses will be performed to describe central tendencies (mean, median) and dispersion (standard deviation, interquartile range) of time to diagnosis. Associations between delay and clinical variables will be explored using regression models.

Expected Outcomes and Relevance:

The investigators anticipate confirming that diagnostic delay is significant in the Brazilian context, similar to international studies. Identifying the stages at which delay occurs (e.g., late presentation, misdiagnosis, referral lag) will allow the design of targeted interventions.

* This study will provide baseline data to support future initiatives such as:
* Educational programs for primary care providers
* Diagnostic algorithms or checklists
* Patient education campaigns
* Policy advocacy for improved rare disease care networks

Ethical Considerations:

This is a non-interventional study involving retrospective review of anonymized patient data. Approval will be obtained from local institutional review boards. No patient consent is required due to the retrospective design.

"This is a mixed observational study including both retrospective and prospective data. Retrospective data will be collected from medical records of patients diagnosed within the past 5 years. In addition, prospective data may be collected during follow-up visits or complementary assessments to complete the diagnostic journey profile, when needed."

ELIGIBILITY:
Inclusion Criteria:

* Availability of documented or estimated date of first symptom suggestive of PAH.
* Availability of documented date of confirmed PAH diagnosis.

Exclusion Criteria:

* Patients with pulmonary hypertension not classified as Group 1 (e.g., due to left heart disease, chronic lung disease, or chronic thromboembolic disease).
* Patients with insufficient data to determine either the date of symptom onset or the date of confirmed diagnosis.
* Patients diagnosed only clinically or by echocardiography, without confirmation by right heart catheterization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with Group 1 Pulmonary Arterial Hypertension (PAH), confirmed by right heart catheterization, who are followed at specialized pulmonary hypertension referral centers in Brazil. Eligible participants must have documented or estimated date of symptom onset and a recorded date of confirmed diagnosis. The study includes patients from diverse geographic regions and healthcare settings to reflect real-world diagnostic practices.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time from Symptom Onset to Confirmed Diagnosis of Group 1 Pulmonary Arterial Hypertension | From date of first reported symptom potentially related to PAH until the date of confirmed diagnosis by right heart catheterization, assessed up to 60 months.
  This outcome measures the time interval (in months) between the patient's first reported symptom potentially related to pulmonary arterial hypertension and the date of confirmed diagnosis by right heart catheterization. Data will be collected through retrospective review of medical records and/or prospectively documented clinical follow-up.

SECONDARY OUTCOMES:
Number of Physicians Consulted Before Diagnosis | From first reported symptom potentially related to PAH until confirmed diagnosis by right heart catheterization, assessed up to 60 months.
  This outcome captures the total number of different physicians (general practitioners and specialists) consulted by the patient between symptom onset and confirmed diagnosis of PAH. This helps identify possible fragmentation or delays in referral.
Number of Misdiagnoses Prior to Final PAH Diagnosis | From first reported symptom potentially related to PAH until confirmed diagnosis by right heart catheterization, assessed up to 60 months.
  This outcome measures how many alternative or incorrect diagnoses the patient received before receiving the definitive diagnosis of PAH. These may include asthma, anxiety, heart failure, or others.
Functional Class at Diagnosis | At baseline (i.e., at the time of confirmed diagnosis by right heart catheterization).
  This outcome records the patient's World Health Organization (WHO) functional class at the time of confirmed diagnosis of PAH. Functional class is a strong prognostic indicator and reflects disease severity at the time of diagnosis.
Time from First Medical Contact to Diagnosis | From first reported symptom potentially related to PAH until confirmed diagnosis by right heart catheterization, assessed up to 60 months.
  This outcome evaluates the delay attributable to the health system by measuring the time (in months) between the patient's first consultation with a healthcare provider and the date of PAH confirmation.

CONTACTS AND LOCATIONS:
Locations (1):
- InCor - Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No